CLINICAL TRIAL: NCT04515849
Title: A Phase 2b, Multicentre, Randomised, Double-blind, Placebo-controlled, and Open-label Comparator Study of Cotadutide in Participants Who Have Chronic Kidney Disease With Type 2 Diabetes Mellitus
Brief Title: A Study of Cotadutide in Participants Who Have Chronic Kidney Disease With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5676C00001; 2020-000255-12 (EudraCT Number)
Record Dates: First submitted 2020-07-06; First posted 2020-08-17 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Diseases
Keywords: MEDI0382; T2DM; Cotadutide; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Diabetic Nephropathies | interventions — cotadutide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cotadutide 100 micrograms (Experimental): Cotadutide 100 micrograms administered subcutaneously
  Interventions: Drug: Cotadutide 100 micrograms
- Cotadutide 300 micrograms (Experimental): Cotadutide 300 micrograms administered subcutaneously
  Interventions: Drug: Cotadutide 300 micrograms
- Cotadutide 600 micrograms (Experimental): Cotadutide 600 micrograms administered subcutaneously
  Interventions: Drug: Cotadutide 600 micrograms
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Drug: Placebo
- Semaglutide (Active Comparator): Semaglutide 1.0 miligrams administered subcutaneously
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Cotadutide 100 micrograms — Cotadutide 100 micrograms administered subcutaneously
  Other Names: MEDI0382
  Arms: Cotadutide 100 micrograms
Drug: Cotadutide 300 micrograms — Cotadutide 300 micrograms administered subcutaneously
  Other Names: MEDI0382
  Arms: Cotadutide 300 micrograms
Drug: Cotadutide 600 micrograms — Cotadutide 600 micrograms administered subcutaneously
  Other Names: MEDI0382
  Arms: Cotadutide 600 micrograms
Drug: Semaglutide — Semaglutide 1.0 miligrams administered subcutaneously
  Other Names: Ozempic
  Arms: Semaglutide
Drug: Placebo — Placebo administered subcutaneously
  Arms: Placebo

SUMMARY:
A Phase 2b, study to measure the effect of Cotadutide at different doses versus placebo or comparator (semaglutide) in participants who have Chronic Kidney Disease with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
A Phase 2b randomised, double-blind, placebo-controlled and open-label active comparator study to evaluate the effect of Cotadutide at 100, 300 or 600 micrograms in participants who have Chronic Kidney Disease with Type 2 Diabetes Mellitus.

The study plans to randomise approximately 225 subjects. Subjects will be randomised to receive double-blind Cotadutide or placebo at 100, 300 or 600 micrograms once daily for 26 weeks, or open-label semaglutide at 1.0 miligrams once a week for 26 weeks. Japanese participants will not be randomised to the semaglutide arm.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate ≥ 20 to < 90 mL/min/1.73 m2 determined at the screening visit or a documented occurrence in medical history at least 3 months prior to randomisation.
* Receiving background standard of care treatment for renal disease and/or T2DM and being treated according to locally recognised guidelines, as appropriate.
* Receiving optimised and stable treatment with an angiotensin-converting-enzyme (ACE) inhibitor or an angiotensin II receptor antagonist for ≥ 3 months at screening at the maximum tolerated dose (MTD) unless contraindicated, not tolerated, or in the opinion of the investigator, not practically available or suitable.
* Micro- or macroalbuminuria as defined by UACR > 50 mg/g or 5.7 mg/mmol.
* Diagnosed with T2DM with glucose control managed with any insulin and/or any oral therapy combination including metformin, SGLT2 inhibitor, thiazolidinedione, or acarbose where no major dose changes (eg, > 50% increase in dose) have occurred within the 4 weeks prior to the start of the run-in period. Participants taking sulfonylureas or glitinides may be randomised following a 4-week washout period of the sulfonylurea/glitinide.
* Haemoglobin A1c range of 6.5 % to 12.5% (inclusive) at screening
* Body mass index > 25 kg/m2 at screening or > 23 kg/m2 for participants enrolled in Japan

Exclusion Criteria:

* History or presence of significant medical or psychological conditions, including significant abnormalities in laboratory parameters or vital signs including ECG, which in the opinion of the investigator, would compromise the participant's safety or successful participation in the study.
* Receiving renal replacement therapy or expected to require it within 6 months of being randomised
* Renal transplant or on the waiting list for renal transplantation
* Received a GLP-1 analogue-containing preparation within the last 30 days or 5 half-lives of the drug, if known (whichever is longer), at the time of Visit 2
* Received any of the following medications within the specified time frame prior to the start of the study (Visit 2):

  1. Aspirin (acetylsalicylic acid) at a dose greater than 150 mg once daily and within the last 3 days prior to the start of the run-in period (Visit 2)
  2. Paracetamol (acetaminophen) or paracetamol-containing preparations at a total daily dose of greater than 3000 mg and within the last 3 days prior to the start of the run-in period (Visit 2)
  3. Ascorbic acid (vitamin C) supplements at a total daily dose of greater than 1000 mg and within the last 3 days prior to the start of the run-in period (Visit 2)
* Participation in another clinical study with an investigational product administered in the last 30 days or 5 half-lives of the drug, if known (whichever is longer)
* Participants with a known severe allergy/hypersensitivity to any of the proposed study interventions or excipients of the product
* Symptoms of acutely decompensated blood glucose control (eg, thirst, polyuria, weight loss) or recent episodes of severe hypoglycaemia
* Type 1 diabetes mellitus (T1DM), history of diabetic ketoacidosis, or clinical suspicion of T1DM
* Participants with recent acute or subacute renal function deterioration
* Significant inflammatory bowel disease, gastroparesis, or other severe disease or surgery affecting the upper gastrointestinal tract (including weight-reducing surgery and procedures) which may affect gastric emptying or could affect the interpretation of safety and tolerability data
* History of acute or chronic pancreatitis
* Significant hepatic disease (except for non-alcoholic steatohepatitis or nonalcoholic fatty liver disease without portal hypertension or cirrhosis) and/or participants with any of the following results:

  1. Aspartate transaminase (AST) ≥ 3 × upper limit of normal (ULN)
  2. Alanine transaminase (ALT) ≥ 3 × ULN
  3. Total bilirubin ≥ 2 × ULN
* Poorly controlled hypertension defined as:

  1. Systolic BP > 180 mm Hg
  2. Diastolic BP ≥ 90 mm Hg after 10 minutes of seated rest and confirmed by repeated measurement at screening. Participants who fail BP screening criteria may be considered for 24-hour ambulatory BP monitoring at the discretion of the investigator. Participants who maintain a mean 24-hour systolic BP ≤ 180 or diastolic BP < 90 mm Hg with a preserved nocturnal dip of > 15% will be considered eligible
* Unstable angina pectoris, myocardial infarction, transient ischemic attack or stroke within 3 months prior to screening, or participants who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 6 months or who are due to undergo these procedures at the time of screening
* Decompensated heart failure or hospitalisation for heart failure in the 3 months prior to screening or symptoms consistent with New York Heart Association heart failure Class III/IV
* Basal calcitonin level > 50 ng/L at screening or history/family history of medullary thyroid carcinoma or multiple endocrine neoplasia
* History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell skin cancer, squamous cell skin cancer, or in situ cervical cancer

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- Australia (9):
  - Research Site, Box Hill
  - Research Site, Elizabeth Vale
  - Research Site, Fitzroy
  - Research Site, Heidelberg
  - Research Site, Melbourne
  - Research Site, Merewether
  - Research Site, Oaklands Park
  - Research Site, Wollongong
  - Research Site, Woolloongabba
- Canada (12):
  - Research Site, Vancouver, British Columbia
  - Research Site, Barrie, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Concord, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
- Germany (12):
  - Research Site, Berlin
  - Research Site, Dortmund
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Kassel
  - Research Site, Ludwigshafen
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Münster
  - Research Site, Riesa
  - Research Site, Sankt Ingbert
- Japan (7):
  - Research Site, Arakawa-ku
  - Research Site, Chitose-shi
  - Research Site, Fujisawa-shi
  - Research Site, Kamakura-shi
  - Research Site, Obihiro-shi
  - Research Site, Sapporo
  - Research Site, Shinjyuku-ku
- New Zealand (7):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Grafton
  - Research Site, Havelock North
  - Research Site, New Plymouth
  - Research Site, Tauranga
  - Research Site, Wellington
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Skierniewice
  - Research Site, Warsaw
  - Research Site, Wierzchosławice
- Spain (14):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Palma
  - Research Site, Palma de Mallorca
  - Research Site, Pozuelo de Alarcón
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Vitoria-Gasteiz
- United Kingdom (3):
  - Research Site, Dundee
  - Research Site, Liverpool
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Result] Selvarajah V, Robertson D, Hansen L, Jermutus L, Smith K, Coggi A, Sanchez J, Chang YT, Yu H, Parkinson J, Khan A, Chung HS, Hess S, Dumas R, Duck T, Jolly S, Elliott TG, Baker J, Lecube A, Derwahl KM, Scott R, Morales C, Peters C, Goldenberg R, Parker VER, Heerspink HJL; study investigators. A randomized phase 2b trial examined the effects of the glucagon-like peptide-1 and glucagon receptor agonist cotadutide on kidney outcomes in patients with diabetic kidney disease. Kidney Int. 2024 Dec;106(6):1170-1180. doi: 10.1016/j.kint.2024.08.023. Epub 2024 Aug 31. PMID 39218393
- [Derived] Yu H, Parker V, Selvarajah V, Hansen L, Robertson D, Hamren B, Khan A, Parkinson J. Pharmacokinetic-pharmacodynamic (PK/PD) modelling of cotadutide effect in patients with chronic kidney disease and type 2 diabetes mellitus. Br J Clin Pharmacol. 2025 Sep;91(9):2672-2683. doi: 10.1002/bcp.70093. Epub 2025 May 9. PMID 40344607
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5676C00001&attachmentIdentifier=6145a98b-b652-4fa3-8311-241cc78fbea6&fileName=CRS_synopsis_redacted.pdf&versionIdentifier=
- See also: CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5676C00001&attachmentIdentifier=bf1fb852-6916-4dbc-b608-5f07c83def73&fileName=CSP_redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5676C00001&attachmentIdentifier=64031a9c-4cab-45ab-8f8d-f2d2427875f3&fileName=SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 79 participating sites in Canada, Australia, New Zealand, Japan, Germany, Poland, Spain and United Kingdom. First subject enrolled 31st August 2020. Last subject last visit: 8th March 2022.
Pre-assignment Details: This is a parallel treatment, double-blind study with 5 arms: Cotadutide 100 mcg,300 mcg&600 mcg,placebo and an open-label semaglutide arm.Outcomes for the cotadutide arms vs. semaglutide were exploratory.Therefore semaglutide arm was excluded from Outcomes.248 patients were enrolled.The study had a 14-day run-in period during which participants followed by a 26-week treatment period and 28-day follow-up period.
Groups:
- Cotadutide 100 ug: Participants randomised to cotadutide 100 µg daily
- Cotadutide 300 ug: Participants randomised to Cotadutide 300 ug daily
- Cotadutide 600 ug: Participants randomised to Cotadutide 600 ug daily
- Placebo ug: Participants randomised to placebo daily
- Semaglutide 1 mg: Participants randomized to semaglutide 1 mg weekly
Period: Overall Study
Arm/Group | Cotadutide 100 ug | Cotadutide 300 ug | Cotadutide 600 ug | Placebo ug | Semaglutide 1 mg
Started | 52 | 49 | 51 | 51 | 45
Completed | 49 | 45 | 50 | 48 | 43
Not Completed | 3 | 4 | 1 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2
Not completed — Death | 2 | 0 | 0 | 0 | 0
Not completed — Other:family emergency | 0 | 0 | 0 | 1 | 0
Not completed — Other:randomised by error | 0 | 1 | 0 | 0 | 0
Not completed — Other:subject hasa to fly to greece for a family emergency and will not be back till 4-5 months | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The numbers above include all participants randomised in the different treatment arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cotadutide 100 ug | Cotadutide 300 ug | Cotadutide 600 ug | Placebo ug | Semaglutide 1 mg | Total
Number analyzed (Participants) | 52 | 49 | 51 | 51 | 45 | 248
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (7.3) | 65.7 (8.8) | 66.1 (7.4) | 69.5 (7.3) | 67.0 (7.8) | 67.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 10 | 13 | 12 | 47
  Male | 43 | 46 | 41 | 38 | 33 | 201
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0 | 0 | 0 | 0
  ASIAN | 10 | 10 | 13 | 10 | 2 | 45
  BLACK OR AFRICAN AMERICAN | 2 | 0 | 0 | 1 | 2 | 5
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 2 | 0 | 1 | 1 | 0 | 4
  OTHER | 0 | 3 | 1 | 0 | 0 | 4
  WHITE | 38 | 36 | 36 | 39 | 41 | 190

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Was Percentage Change in UACR of Cotadutide at Different Dose Levels Compared to Placebo After 14 Weeks
Description: Percentage change in UACR of cotadutide at different dose levels compared to placebo after 14 weeks. Efficacy endpoints for cotadutide vs. semaglutide are exploratory and are therefore excluded.
Time Frame: Baseline to the end of 14 weeks of dosing
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percentage change
Groups:
- Cotadutide 300 µg: Participants randomised to cotadutide 300 µg
- Cotadutide 600 µg: Participants randomised to cotadutide 600 µg
Arm/Group | Cotadutide 100 ug | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 49 | 43 | 37 | 43
Percentage change | -10.96 [-29.60 to 12.61] | -40.47 [-53.00 to -24.60] | -44.60 [-56.21 to -29.91] | 4.60 [-18.02 to 33.46]

2. Secondary Outcome: Percentage Change in UACR of Cotadutide at Different Dose Levels Compared to Placebo After 26 Weeks
Description: Percentage change in UACR of cotadutide at different dose levels compared to placebo from baseline to end of 26 weeks. Efficacy endpoints for cotadutide vs. semaglutide are exploratory and are therefore excluded.
Time Frame: Baseline to end of 26 weeks of dosing
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percentage change
Groups:
- Cotadutide 600 µg: Number of participants randomised to cotadutide 600 µg
Arm/Group | Cotadutide 100 ug | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 49 | 46 | 48 | 49
Percentage change | -17.85 [-45.47 to 23.78] | -38.68 [-59.61 to -6.88] | -57.87 [-73.33 to -33.45] | 11.79 [-27.85 to 73.22]

3. Secondary Outcome: Percent Change in Body Weight of Cotatudide at Different Dose Levels Versus Placebo From Baseline to End of 14 Weeks of Dosing
Description: Percentage change in body weight of cotadutide at different dose levels compared to placebo from baseline to end of 14 weeks of dosing.
Time Frame: Baseline to end of 14 weeks of dosing
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Cotadutide 100 ug | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 37 | 32 | 27 | 35
Percentage change | -2.84 (0.65) | -4.15 (0.68) | -5.40 (0.73) | -1.61 (0.66)

4. Secondary Outcome: Percentage Change in Body Weight of Cotadutide at Different Dose Levels Versus Placebo From Baseline to End of 26 Weeks of Dosing
Description: Percentage change in body weight of cotadutide at different dose levels compared to placebo from baseline to end of 26 weeks of dosing
Time Frame: Baseline to end of 26 weeks of dosing
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Cotadutide 100 ug | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 37 | 33 | 27 | 35
Percentage change | -2.60 (0.89) | -5.45 (0.92) | -7.35 (0.99) | -2.23 (0.90)

5. Secondary Outcome: Percent Change in HbA1c of Cotadutide at Different Dose Levels Versus Placebo From Baseline to the End of 14 of Dosing
Description: Percentage change in HbA1c of cotadutide at different dose levels compared to placebo from baseline to end of 14 weeks of dosing
Time Frame: Baseline to end of 14 weeks of dosing
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Cotadutide 100 µg: Participants randomised to Cotadutide 100 µg
Arm/Group | Cotadutide 100 µg | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 49 | 45 | 48 | 39
Percent change | -0.76 (0.12) | -0.82 (0.12) | -0.65 (0.12) | -0.08 (0.12)

6. Secondary Outcome: Percent Change in HbA1c of Cotadutide at Different Dose Levels Versus Placebo From Baseline to the End of 26 of Dosing
Description: Percentage change in HbA1c of cotadutide at different dose levels compared to placebo from baseline to end of 26 weeks of dosing
Time Frame: Baseline to end of 26 weeks of dosing
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Cotadutide 100 µg | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 49 | 46 | 48 | 39
Percent change | -0.92 (0.11) | -0.92 (0.11) | -0.89 (0.11) | -0.25 (0.11)

7. Secondary Outcome: Change in Fasting Glucose of Cotadutide at Different Dose Levels From Baseline Versus Placebo After 14 Weeks of Dosing
Description: Absolute change in fasting glucose of cotadutide at different dose levels compared to placebo from baseline to end of 14 weeks
Time Frame: Baseline to end of 14 weeks of dosing
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Cotadutide 100 ug | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 42 | 45 | 48 | 49
mmol/L | -1.35 (0.37) | -1.57 (0.35) | -1.69 (0.40) | -0.54 (0.37)

8. Secondary Outcome: Change in Fasting Glucose of Cotadutide at Different Dose Levels From Baseline Versus Placebo After 26 Weeks of Dosing
Description: Absolute change in fasting glucose of cotadutide at different dose levels compared to placebo from baseline to end of 26 weeks
Time Frame: Baseline to end of 26 weeks of dosing
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Cotadutide 100 ug | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 45 | 43 | 39 | 45
mmol/L | -1.78 (0.36) | -1.76 (0.37) | -1.57 (0.39) | -0.72 (0.37)

9. Secondary Outcome: Change in 10-day Average Glucose Levels of Cotadutide at Different Dose Levels Versus Placebo From Baseline to End of 14 Weeks of Dosing
Description: Absolute change in 10-day average glucose of cotadutide at different dose levels compared to placebo from baseline to end of 14 weeks of dosing
Time Frame: Baseline to end of 14 weeks of dosing
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Cotadutide 100 ug | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 30 | 25 | 26 | 30
mmol/L | -1.556 (0.320) | -1.478 (0.337) | -1.269 (0.334) | -0.440 (0.311)

10. Secondary Outcome: Change in 10-day Average Glucose Levels of Cotadutide at Different Dose Levels Versus Placebo From Baseline to End of 26 Weeks of Dosing
Description: Absolute change in 10-day average glucose of cotadutide at different dose levels compared to placebo from baseline to end of 26 weeks of dosing
Time Frame: Baseline to end of 26 weeks of dosing
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Cotadutide 100 ug | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 25 | 18 | 22 | 30
mmol/L | -1.735 (0.307) | -1.446 (0.334) | -1.118 (0.321) | -0.273 (0.290)

11. Secondary Outcome: Change in Percentage Time Spent in Hyperglycaemia Over 10 Days of Cotadutide at Different Dose Levels Compared to Placebo After 14 Weeks of Dosing
Description: Percentage change in 10-day percentage time spent in hyperglycaemia of cotadutide at different dose levels compared to placebo from baseline to end of 14 weeks
Time Frame: Baseline to 14 weeks of dosing
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Cotadutide 100 ug | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 30 | 25 | 26 | 30
Percent Change | -13.87 (3.35) | -15.79 (3.55) | -13.90 (3.52) | -4.09 (3.27)

12. Secondary Outcome: Change in Percentage Time Spent in Hyperglycaemia Over 10 Days of Cotadutide at Different Dose Levels Compared to Placebo After 26 Weeks of Dosing
Description: Percentage change in 10-day percentage time spent in hyperglycaemia of cotadutide at different dose levels compared to placebo from baseline to end of 26 weeks
Time Frame: Baseline to 26 weeks of dosing
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Cotadutide 100 ug | Cotadutide 300 µg | Cotadutide 600 µg | Placebo ug
Number analyzed (Participants) | 25 | 18 | 22 | 27
Percent change | -18.06 (3.33) | -15.38 (3.76) | -11.91 (3.51) | -3.00 (3.17)

ADVERSE EVENTS:
Time Frame: Screening throughout the treatment period and including the follow-up period (28 days post last dose), an average of 37 weeks.
Arm/Group | Cotadutide 100 ug | Cotadutide 300 ug | Cotadutide 600 ug | Placebo ug | Semaglutide 1 mg
All-Cause Mortality (participants affected / at risk) | 2/52 | 0/49 | 0/51 | 0/51 | 0/45
Serious Adverse Events (participants affected / at risk) | 5/52 | 5/49 | 5/51 | 5/51 | 5/45
Other Adverse Events (participants affected / at risk) | 43/52 | 38/49 | 38/51 | 38/51 | 39/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cotadutide 100 ug (N=52) | Cotadutide 300 ug (N=49) | Cotadutide 600 ug (N=51) | Placebo ug (N=51) | Semaglutide 1 mg (N=45)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder with anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suspected suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cotadutide 100 ug (N=52) | Cotadutide 300 ug (N=49) | Cotadutide 600 ug (N=51) | Placebo ug (N=51) | Semaglutide 1 mg (N=45)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Costal cartilage fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin pressure mark (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Blood bicarbonate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pedal pulse decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary arterial pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulse absent (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine output increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular internal diameter (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 8 (8)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0/0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 13 (88) | 16 (106) | 13 (83) | 13 (148) | 4 (4)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0/45 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Akinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (5) | 1 (2) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7) | 2 (3) | 5 (7) | 2 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 7 (10) | 6 (9) | 4 (8) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 7 (9) | 14 (18) | 5 (5) | 12 (12)
Oral lichen planus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 7 (12) | 2 (2) | 7 (7)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 1 (2) | 2 (2)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac septal hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lichenification (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Meniscus removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 5 (5)
Asymptomatic covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT04515849/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT04515849/SAP_001.pdf